CLINICAL TRIAL: NCT05471817
Title: Open-label, Fixed Sequence Crossover Study to Determine the Effects of a Single Dose of Elinzanetant (BAY 3427080) on the Pharmacokinetics of Dabigatran Etexilate in Healthy Participants
Brief Title: A Study to Learn How the Study Drug Elinzanetant (BAY 3427080) Affects the Way the Drug Dabigatran Moves Into, Through and Out of the Body in Healthy Male and Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 22081; 2022-500201-41-00 (Other: EU CT Number)
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Vasomotor Symptoms as a Sex Hormone-dependent Disorder in Women and Men; Hot Flashes; Healthy Volunteers
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Hot Flashes | interventions — Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EZN - DBG (Experimental): Participants will receive a single oral dose of dabigatran (DBG) etexilate in fasted state in Period 1; followed by a single oral dose of elinzanetant (EZN) and DBG etexilate (30 min after EZN) in fasted state in Period 2.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Dabigatran etexilate

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) — Capsule, oral, single dose
Drug: Dabigatran etexilate — Capsule, oral, single dose
  Other Names: Pradaxa

SUMMARY:
Researchers are looking for a better way to treat men and women with vasomotor symptoms, a condition of having hot flashes caused by hormonal changes.

The study drug, elinzanetant, is under development to treat symptoms caused by hormonal changes. It works by blocking a substance called neurokinin from sending signals to other parts of the body, which is thought to play a role in starting hot flashes.

Participants of this study will be healthy and will have no benefit from administration of elinzanetant. This study, however, will provide information on how to use elinzanetant in people with vasomotor symptoms.

The main purpose of this study is to learn whether the study drug elinzanetant (BAY3427080) affects the way the substrate drug dabigatran moves into, through and out of the body.

One way of removing substances such as drugs from the body are proteins which act as transporters. One such transporter is called P-gp. As a so-called substrate of P-gp, dabigatran is typically removed from the body by P-gp transporters.

The activity of transporters can be increased by substances called inducers and decreased by substances called inhibitors. It has been found in laboratory experiments that the study drug elinzanetant is a weak inhibitor of the P-gp transporter. Inhibition of this transporter can lead to an increase in the amount of drugs such as dabigatran in the blood.

This study is therefore needed to make recommendations on how elinzanetant can be used safely together with other drugs that are removed from the body by the P-gp transporter.

To answer this, the researchers will compare

* the average highest level of dabigatran in the blood (also referred to as Cmax)
* the average total level of dabigatran in the blood (also referred to as AUC) when dabigatran is given alone and is given together with elinzanetant. All participants will take one dose of dabigatran by mouth in the first period of the study. And after 4 days, the participants will take one dose of elinzanetant by mouth and at 30 minutes later, one dose of dabigatran by mouth during the second period of the study. The total duration of individual study participation will be about 4.5 weeks including the screening period. Each participant will stay in the center for 9 days with 8 overnight stays.

During the study, the study team will:

* take blood and urine samples
* do physical examinations
* check the participants' overall health
* examine heart health using ECG
* check vital signs
* ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, blood pressure (BP), pulse rate, 12-lead electrocardiogram (ECG), and laboratory tests.
* Body weight of at least 50 kg and body mass index (BMI) above or equal 18.0 and below or equal 30.0 kg/m² at screening.
* Male or female
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Known hypersensitivity to any study intervention (active substances or excipients of the preparations) to be used in the study.
* Thyroid-stimulating hormone (TSH) outside normal range at screening.
* Any lesion or condition considered a significant risk factor for major bleeding.
* Known or suspected coagulopathies.
* Estimated glomerular filtration rate (eGFR according to Chronic Kidney Disease Epidemiology Collaboration; CKD-EPI) below 90 mL/min/1.73 m2 at screening.
* Any use of systemic or topically active medication or herbal remedies, prescription or non-prescription, within 2 weeks or 5 half-lives (whichever longer) prior to the first study intervention administration.
* Suspicion of drug or alcohol abuse.
* Smoker (current, or within 6 months before screening).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Cmax of unconjugated and total dabigatran when given without or together with a single oral dose of elinzanetant | Pre-dose and up until 72 hours post-dose of DBG etexilate
  Cmax: maximum observed drug concentration in plasma after single dose
AUC of unconjugated and total dabigatran when given without or together with a single oral dose of elinzanetant | Pre-dose and up until 72 hours post-dose of DBG etexilate
  AUC(0-tlast) will be the primary endpoint if AUC cannot be determined in all participants. AUC: area under the concentration vs. time curve from zero to infinity after single dose; AUC(0-tlast): area under the concentration vs. time curve from zero to last quantifiable concentration after single dose

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | After first study intervention in Period 1 and up to 72.5 hours post-dose of elinzanetant in Period 2 (around 8 days)
Number of participants with treatment-emergent adverse events (TEAEs) categorized by severity | After first study intervention in Period 1 and up to 72.5 hours post-dose of elinzanetant in Period 2 (around 8 days)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Wuppertal GmbH, Wuppertal, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.